CLINICAL TRIAL: NCT03759028
Title: A Randomized Controlled Trial of Acetaminophen and Ibuprofen Versus Acetaminophen and Oxycodone for Postoperative Pain Control in Operative Pediatric Supracondylar Humerus Fracture
Brief Title: Supracondylar Post-Operative Pain Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mauricio Silva, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB# 18-001158
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Supracondylar Humerus Fracture
Keywords: closed reduction percutaneous pinning; post-operative pain control; opioid; pediatric; elbow fracture
MeSH Terms: conditions — Elbow Fractures | interventions — Ibuprofen; Oxycodone; Acetaminophen

STUDY DESIGN:
Intervention Model Description: double blinded, randomized trial
Who Masked: Participant, Investigator
Masking Description: Randomization envelopes used to allocate treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ibuprofen (Experimental): This group is given acetaminophen (liquid oral medication, 15mg/kg/dose every 6 hours as needed, max 90mg/kg/day) as the first-line pain medication, and as needed ibuprofen for breakthrough pain (liquid oral medication, 10mg/kg/dose every 8 hours as needed, max dose 40mg/kg/day).
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen
- Oxycodone (Active Comparator): This group is given acetaminophen (liquid oral medication, 15mg/kg/dose every 6 hours as needed, max 90mg/kg/day) as the first-line pain medication, and as needed oxycodone for breakthrough pain (liquid oral medication, 0.1mg/kg/dose every 6 hours as needed).
  Interventions: Drug: Oxycodone; Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — Post-operative pain control protocol of closed reduction percutaneous pinning of supracondylar humerus fracture.
  Other Names: Advil, Motrin
  Arms: Ibuprofen
Drug: Oxycodone — Post-operative pain control protocol of closed reduction percutaneous pinning of supracondylar humerus fracture.
  Other Names: roxicodone
  Arms: Oxycodone
Drug: Acetaminophen — Post-operative pain control protocol of closed reduction percutaneous pinning of supracondylar humerus fracture.
  Other Names: Tylenol, Paracetamol

SUMMARY:
The purpose of this study to investigate post-operative pain control in pediatric patients with closed supracondylar humerus fracture who undergo closed reduction and percutaneous pinning. Currently, it is standard of care that patients receive a narcotic prescription for post-operative pain control. All patients will initially be seen in our pediatric urgent care and recruited at the time of surgery. Patients will be randomized to receiving acetaminophen and ibuprofen or acetaminophen and oxycodone. Parents will not be blinded to the acetaminophen but both investigators, parents and the patients will be blinded to the study drug (ibuprofen or oxycodone). Pain level will be assessed using the Wong-Baker FACES scale and parents will be asked to fill out a questionnaire regarding their satisfaction with the surgery and pain control. Parents will also fill out a medication log until the patient no longer requires pain medication. The duration of participation in the study is approximately 1 week and requires 2 visits (time of recruitment at surgery to 1st post-op visit). This study is being conducted in hopes of reducing opioid prescription after surgical fixation of uncomplicated supracondylar humerus fractures if our study can show that patient's pain levels post-operatively and parent/patient satisfaction are unchanged or improved in the acetaminophen and ibuprofen arm.

DETAILED DESCRIPTION:
This is a double-blinded, randomized controlled trial comparing the analgesic efficacy between acetaminophen and ibuprofen versus acetaminophen and oxycodone for postoperative pain control in patients following closed reduction and percutaneous pinning for isolated closed supracondylar humerus fractures. Each patient will be evaluated initially at our institution's pediatric urgent care center and placed in a long arm splint with instructions to elevate the affected arm. Patients will not be discharged with any prescriptions for narcotic pain medication and will be instructed to take weight-based doses of acetaminophen and/or ibuprofen for pain control as needed.

All patients age 5-12 with closed Gartland type II supracondylar humerus fractures requiring fixation (e.g. satisfactory reduction not achieved with closed reduction and casting or medial column comminution) and Gartland type III supracondylar humerus fractures scheduled for surgery will be approached for participation in the study. Demographic data (age, gender, weight, height, ethnicity, primary language spoken at home, insurance type) will be obtained through chart review on each included patient.

The exclusion criteria include open fractures, fractures with concomitant vascular or neurologic deficit, any fracture requiring open reduction, pathologic fractures, those presenting with concomitant injuries, swelling requiring post-operative hospitalization for monitoring, any known history of allergies to acetaminophen, ibuprofen or oxycodone, and patients with developmental delay that would preclude participation in the visual analog Faces Pain Scale-Revised. Informed consent will be obtained from all parents who wish to participate in the study, and assent will be obtained from patients when possible. If parents refuse participation in the study, the reason for refusal will be documented, and their child's care and post-operative protocol will be consistent with our typical protocol, which includes all 3 medications.

All surgeries will be performed at our outpatient surgery center. The treating pediatric anesthesiologists will use a standardized anesthesia protocol. All patients will be under general anesthesia and will not receive any regional anesthetics or local anesthetics. All included patients will undergo closed reduction and percutaneous pinning using 2-3 pins placed either all laterally or medially and laterally by two pediatric orthopaedic surgeons (MS and RT). They will al be placed in posterior long arm splints thereafter and made non-weight bearing in that extremity. The patients will be transferred to our post-anesthesia care unit (PACU), where morphine IV 0.1mg/kg will be utilized as needed for before discharge home. Nursing staff will record the amount of pain medication provided in the PACU as well as the pre-discharge pain scores, as is our typical post-operative protocol.

Prior to discharge, patients will be randomized to receiving acetaminophen for first-line medication (liquid oral medication, 15mg/kg/dose every 6 hours as needed, max 90mg/kg/day) with as needed ibuprofen for breakthrough pain (liquid oral medication, 10mg/kg/dose every 8 hours as needed, max dose 40mg/kg/day) or acetaminophen for first-line medication (liquid oral medication, 15mg/kg/dose every 6 hours as needed, max 90mg/kg/day) with as needed oxycodone for breakthrough pain (liquid oral medication, 0.1mg/kg/dose every 6 hours as needed). Each patient will receive 18 doses (3 days) of acetaminophen and the study medication. Pre-sealed, sequentially numbered randomization envelopes containing each subject's group will be delivered to the hospital pharmacy. Patients will be instructed to first take the labeled acetaminophen medication and to take the study medication (unlabeled) as needed for breakthrough pain as prescribed. Patients will be given both patient information for both study medications in order to keep the patients blinded to which study medication they received. They will be given patient information for both medications but told that they have been given only one of the two medications. Medication labels will be obscured by the pharmacist with a circumferential tape. Throughout the study, the investigators and the parents will be blinded as to which study medication was given to each participant. Parents who contact the physician (a resident physician on-call for the pediatric orthopaedic surgery service who is not involved in the study) post-operatively for alternative pain medication will be provided the study medication not initially provided (i.e. those that were randomized to receive oxycodone primarily will be provided ibuprofen and vice versa), as confirmed by our pharmacy.

Post-operatively, the parents of each participant will be asked to use the Faces Pain Scale-Revised (FPS-R)16 to rate the child's level of pain at 24 hours and 48 hours after surgery. A research team member will call each participant's guardian at 24 and 48 hours post-operatively to collect these responses. Parents will further be asked to complete the modified Total Quality Pain Management Instrument (TQPM)17 regarding their level of satisfaction with surgery and post-operative pain control. Parents will be asked to report any side effects (e.g. nausea, vomiting, lethargy, constipation) associated with the medications. A take-home medication log will be utilized by the parents to record the type and amount of mediation given to each participant and to record any associated side effects.

For breakthrough pain experienced during pharmacy hours the patient will have the option to return to our pharmacy to obtain the medication they were not originally prescribed. Though the investigators believe this will be unlikely, if they are unable to get to the pharmacy for the other medication (e.g. oxycodone if they were in the ibuprofen group or ibuprofen if they were in the oxycodone group), parents can go to the ER for IM/IV medication for pain relief and they can get a prescription for oxycodone or ibuprofen from the ER if necessary, once they contact the resident on call. There will always be a resident on call 24/7 to advise patients if they are unable to achieve adequate pain control with medications received. Again, the study group believes this will be an unlikely/rare event. The resident on call will have access to the study medication that the patient received. At this point, the resident on call can reveal what medication they were getting (in case they need a new prescription from the ER) so they do not get oxycodone if they were already prescribed oxycodone (and can get something different) or they have the option to obtain ibuprofen over-the-counter if they wish. Patients who need to get the other medication would be considered a "failure in treatment" and would not be analyzed together from the original group.

ELIGIBILITY:
Inclusion Criteria:

* Closed supracondylar humerus fracture
* Isolated supracondylar humerus fracture
* Type II and III supracondylar humerus fracture
* Fractures treated with closed reduction percutaneous pinning

Exclusion Criteria:

* Fractures with concomitant vascular injury
* Fractures with concomitant neurologic deficit
* Pathologic fractures
* Fractures with concomitant injuries (multiple trauma)
* Fractures with swelling requiring post-operative hospitalization for monitoring
* Known history of allergies to acetaminophen, ibuprofen or oxycodone
* Patients with developmental delay that would preclude participation in the visual analog Faces Pain Scale-Revised
* Patients with intellectual disability that would preclude participation in the visual analog Faces Pain Scale-Revised
* History of suspected child abuse

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Faces Pain Scale-Revised (FPSR) | 24 to 48 hours post-operatively
  Self reported measure of pain on scale 0-10. 0 = no pain; 10 = worst pain imaginable

SECONDARY OUTCOMES:
Total Quality Pain Management Instrument | 1 week at first post-operative follow-up
  Questionnaire used to measure the quality of children's post-operative pain management in which parents and patients are asked multiple questions re: post-operative pain management including domains in pain experience, pain relief, adverse effects, future analgesic use. The majority of the questions are binary, but there are a few questions that include a mild, moderate, severe option. There is no numerical output, and the subscales are not combined.

OTHER OUTCOMES:
Pain medication logs | Immediately after surgery at time of randomization until the patient returns for 1st post-operative visit, 7-10 days post-operatively, assessed up to 10 days.
  Self report take home medication logs recording the time, type, dosage, and side effects of medication

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Silva, MD, Principal Investigator — UCLA/OIC
Locations (1):
- Orthopaedic Institute for Children, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03759028/Prot_005.pdf
  • Informed Consent Form: Parent Consent SCHF Pain (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03759028/ICF_003.pdf
  • Informed Consent Form: Child Assent SCHF Pain (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03759028/ICF_004.pdf